CLINICAL TRIAL: NCT05708703
Title: Time Toxicity of Cancer: the Time Demands of Cancer-related Activities and Their Impact on Well-being and Quality of Life
Brief Title: Assessing the Time Demands of Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2022LS100; 1R01CA277714-01 (NIH)
Record Dates: First submitted 2023-01-20; First posted 2023-02-01 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer; Ovarian Cancer
Keywords: ovarian cancer; metastatic breast cancer; time use; quality of life; cancer survivorship
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Individuals receiving treatment for metastatic breast cancer or advanced stage ovarian cancer, will complete a baseline survey, install a mobile app on their smartphone to track daily activities, short daily surveys, and a study end survey

SUMMARY:
A total of 80 individuals receiving treatment for metastatic breast or advanced stage ovarian cancer will be asked to complete a baseline survey and install the mobile app on their smartphone; carry the smartphone for 28 consecutive days while outside the home; keep smartphone location and motion services active; confirm and correct (if needed) smartphone-detected activities and trips; use the app interface to provide additional information on activities and trips related to cancer treatment tasks; complete daily surveys regarding well-being; and at the end of the 28 day period, complete an online survey.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with advanced stage (III, IV) ovarian (ovarian, fallopian tube or primary peritoneal) or metastatic breast cancer [do not need to be newly diagnosed]
* Currently receiving any type of therapy for their cancer [can be front-line, maintenance therapy, or treatment for recurrence]
* Able to complete study tasks in English
* Able to provide voluntary informed consent
* Own an Android or iOS smartphone on which the operating system is version 9.0 or higher for Android or 10.0 higher for iOS; or willing to use a researcher-provided smartphone

Exclusion Criteria:

* Those who are currently incarcerated
* Have opted out of research contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is for patients with either breast or ovarian cancer.
Study Population: Individuals currently undergoing treatment for metastatic breast or advanced stage ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2030-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Vogel, Ph.D., Principal Investigator — University of Minnesota Masonic Cancer Center
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - Masonic Cancer Center - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
The following data (for which we will obtain participant consent to share in de-identified form) will be collected as part of the project and will be available for sharing in raw or aggregate form. Specifically, any individual level data will be de-identified before sharing. Demographic data may only be shared at an aggregated level as needed to maintain confidentiality.
  * Survey data (baseline, day 28)
  * Mobile application activity and well-being data
  The data will be archived and shared and the University of Minnesota Libraries will serve as the steward of the de-identified, archived dataset from that point forward.
Time Frame: Data will deposited into the repository as soon as possible but no later than within one year of the completion of the funded project period or upon acceptance of the data for publication, whichever is earlier.
Access Criteria: The de-identified data will be available to all interested parties. No specific data sharing agreement will be needed for DRUM; however, DRUM does have a general end-user access policy available online.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Cohort
Started | 78
Completed | 60
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Study Cohort
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 59
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Time Spent on Cancer-related Care Tasks at Home
Description: Summary of mobile app smartphone collected data from daily surveys about time spent at home on cancer-related care tasks over 28 days, including taking medications, scheduling appointments, handling medical bills, managing symptoms, monitoring health status and arranging help/transportation.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: minutes per week
Arm/Group | Study Cohort
Number analyzed (Participants) | 60
minutes per week | 196 [116 to 321]

2. Primary Outcome: Time Spent on All Cancer-related Care Tasks (Out-of-home and at Home)
Description: Summary of mobile app smartphone collected data from daily trips and surveys about time spent at home on cancer-related care tasks over 28 days, including out-of-home healthcare encounters, travel time, and at-home tasks including taking medications, scheduling appointments, handling medical bills, managing symptoms, monitoring health status and arranging help/transportation.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: minutes per week
Arm/Group | Study Cohort
Number analyzed (Participants) | 60
minutes per week | 404 [265 to 599]

3. Primary Outcome: Out-of-home Cancer-related Healthcare Encounters
Description: Summary of mobile app smartphone collected from daily-recorded trips away from home, collected over 28 days, focusing on those denoted as being related to cancer care (e.g. clinic visit, treatment, lab, pharmacy, imaging).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: episodes per month
Arm/Group | Study Cohort
Number analyzed (Participants) | 60
episodes per month | 4.9 (3.1)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT05708703/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT05708703/ICF_001.pdf